CLINICAL TRIAL: NCT07055438
Title: Analgesic Efficacy of Ultrasound Guided Bilateral External Oblique Intercostal Plane Block Versus Rectus Sheath Block in Upper Abdominal Surgeries: A Randomized Double-blinded Controlled Study
Brief Title: Bilateral External Oblique Intercostal Plane Bock (EOIPB) in Upper Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Associate professor of Anesthesia, intesive care and pain management - Kasr El Aini Hospital, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-185-2024
Record Dates: First submitted 2025-06-15; First posted 2025-07-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Analgesia
Keywords: Rectus shealth block; External oblique intercostal plane block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSB (Active Comparator): Bilateral rectus sheath block for patients undergoing upper abdominal surgeries
  Interventions: Procedure: Ultrasound guided Rectus sheath block
- EOIPB (Experimental): Bilateral External oblique intercostal plane block for patients undergoing upper abdominal surgeries
  Interventions: Procedure: ultrasound guided external oblique intercostal plane block

INTERVENTIONS:
Procedure: Ultrasound guided Rectus sheath block — After receiving general anesthesia, bilateral ultrasound guided rectus sheath block with 20 ml of 0.25% bupivacaine on each side will be administered to 20 patients undergoing upper abdominal surgeries namely whipple operation and total gastrectomy
  Arms: RSB
Procedure: ultrasound guided external oblique intercostal plane block — After receiving general anesthesia, bilateral ultrasound guided external oblique intercostal plane block with 20 ml of 0.25% bupivacaine on each side will be administered to 20 patients undergoing upper abdominal surgeries namely whipple operation and total gastrectomy
  Arms: EOIPB

SUMMARY:
The current study is designed to investigate the analgesic potentials of two modalities of abdominal blocks where local anesthetics is injected in the fascial planes of the abdominal muscles to anesthetize the nerves supplying the abdomen in patients undergoing upper abdomial surgeries.

the two modalities are the rectus sheath block (RSB) and the external oblique intercostal plane block (EOIPB). The investigators are going to use the ultrasound to identify the muscles and inject the local anesthetics. The investigators suggest that the EOIPB might provide better pain control when compared to RSB.

DETAILED DESCRIPTION:
Fascial plane blocks emerge as an appealing technique to provide good intraoperative and postoperative analgesia in patients undergoing upper abdominal surgeries. Such techniques have the benefit of decreasing opioids use and consequently reducing the like hood of their side effects.

Ultrasound guided rectus sheath Block (RSB) targets the terminal branches of thoracic nerves thus providing analgesia for midline abdominal incisions.

Ultrasound guided external oblique intercostal plane block (EOIPB), a relatively new technique, targets the lateral cutaneous branches of the thoracoabdominal nerves providing analgesia for anterolateral and upper median plane of the abdomen.

Studies Comparing both techniques are deficient, that is why the investigators designed the current study to evaluate and compare the analgesic efficacy of both techniques in upper abdominal surgeries namely Whipple operation and total gastrectomy.

The study is a randomized controlled double blinded trial comprising two groups. The RSB group will receive bilateral ultrasound guided rectus sheath block with 20ml of 0.25% bupivacaine on each side. The EOIB group will receive bilateral ultrasound guided External oblique intercostal plane block with 20ml of 0.25% bupivacaine on each side as well. Both blocks will be performed after administering general anesthesia.

The main endpoint of the study is the time to first request for rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 Years
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status II, III.
* Patients who will undergo upper abdominal surgeries (Whipple operation, total gastrectomy).

Exclusion Criteria:

* Coagulation disorders.
* Abdominal surgery history.
* Infection in the block application area.
* Chronic opioid use.
* Local anesthetic (LA) allergy.
* Pregnancy.
* BMI ≥35 kg/m2.
* Severe cardiovascular problems.
* Diabetic neuropathy.
* Complicated surgeries with massive blood loss and hemodynamic instability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-24 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Time to first request for rescue analgesia | Time in hours from end of surgery to first dose of morphine administered up to 24 hours postoperatively
  Time from end of surgery to first dose of morphine administered

SECONDARY OUTCOMES:
Fentanyl consumption | From the start of the surgery till the end in micogram/Kg
  Intraoperative fentanyl consumption
Postoperative morphine consumption | from the time numerical rating scale exceeds 3 and till 24 hours after the end of the surgery
  Total morphine consumption (mg) in the first 24hrs after surgery
Pain score | from the time of recovery immediately in the postoperative period and then at 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 12 hours and 24 hours postoperatively
  Pain score using Numerical rating Scale (NRS)between 0 and 10, Zero means no pain and ten means the worst pain
Patient satisfaction of analgesia | 2 hours after recovery from anesthesia
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied ; 5, extremely satisfied)
Incidence of postoperative nausea and vomiting | From the recovery of anesthesia and up to 24 hours postoperatively
  The number of patients suffering from postoperative nausea and vomiting in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd El Fattah, Associate professor, Principal Investigator — National Cancer Institute, Egypt
Locations (2):
- Egypt (2):
  - Kasr El Ainy, Cairo
  - National Cancer institute, Cairo

IPD SHARING:
Plan to Share IPD: Yes
The detailed protocol describing the techniques used in the study and the anesthetic conduct and the outcome measures.
  The statistical plan to analyze the different outcome measures.
Supporting Information: Study Protocol, SAP
Time Frame: IPD can be available 2 months after completion of the study
Access Criteria: IPD can be accessed from the authors by journals considering the study for publication and upon reasonable request from other investigators

REFERENCES:
- [Result] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112
- [Result] Ohgoshi Y, Kawagoe I, Ando A, Ikegami M, Hanai S, Ichimura K. Novel external oblique muscle plane block for blockade of the lateral abdominal wall: a pilot study on volunteers. Can J Anaesth. 2022 Oct;69(10):1203-1210. doi: 10.1007/s12630-022-02310-4. Epub 2022 Aug 23. PMID 35999334
- [Result] Abdildin Y, Tapinova K, Salamat A, Shaimakhanov R, Aitbayev A, Viderman D. Rectus Sheath Block in Abdominal Surgery: A Systematic Review with Meta-Analysis. Rom J Anaesth Intensive Care. 2023 Apr 20;30(1):43-50. doi: 10.2478/rjaic-2023-0006. eCollection 2023 Apr. PMID 37635853
- [Result] Cho S, Kim YJ, Jeong K, Moon HS. Ultrasound-guided bilateral rectus sheath block reduces early postoperative pain after laparoscopic gynecologic surgery: a randomized study. J Anesth. 2018 Apr;32(2):189-197. doi: 10.1007/s00540-018-2457-0. Epub 2018 Feb 8. PMID 29423579
- [Result] Howle R, Ng SC, Wong HY, Onwochei D, Desai N. Comparison of analgesic modalities for patients undergoing midline laparotomy: a systematic review and network meta-analysis. Can J Anaesth. 2022 Jan;69(1):140-176. doi: 10.1007/s12630-021-02128-6. Epub 2021 Nov 5. PMID 34739706